CLINICAL TRIAL: NCT04097509
Title: Comparison of the Effects of Different Platelet Concentrates on Palatal Wound Healing
Brief Title: Effects of Platelet Concentrates on Palatal Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, mustafa özay uslu, Assistant professor, Faculty of Dentistry, Department of Periodontology, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018/46
Record Dates: First submitted 2019-09-17; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Wound Heal; Platelets; Defect; Periodontal Inflammation; Gingival Recession
MeSH Terms: conditions — Blood Platelet Disorders; Gingival Recession

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized, controlled clinical trial. Three groups were randomly assigned as one control and two test groups. A total of 36 patients (12 patients in each group) were included in the study. In the control group, only moist sterile tamponade was applied following graft removal to the palatinal donor area. In the test groups, polymerized AFG or polymerized i-PRF were applied to the donor area. After these procedures, donor palate was closed with sterile aluminum foil and periodontal pat in all 3 groups.
Who Masked: Participant, Investigator
Masking Description: The patient and investigator were blinded to the applications
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- autologous fibrin glue (AFG) group (Experimental): In the test groups, polymerized AFG was applied to the palatinal donor area. Donor palate was closed with sterile aluminum foil and periodontal pack
  Interventions: Biological: AFG application on palatinal wound healing
- injectable platelet rich fibrin (i-PRF) group (Experimental): In the test groups, polymerized i-PRF was applied to the donor area. Donor palate was closed with sterile aluminum foil and periodontal pack.
  Interventions: Biological: i-PRF application on palatinal wound healing
- Control Group (Placebo Comparator): In the control group, only moist sterile tamponade was applied following graft removal to the palatinal donor area. Donor palate was closed with sterile aluminum foil and periodontal pack
  Interventions: Other: control

INTERVENTIONS:
Biological: AFG application on palatinal wound healing — 9 ml venous blood collected from the patient was transferred to the tube without any anticoagulants. In the protocol, venous blood collected in the tube was centrifuged for 2 minutes at 2700 rpm (approximately 692 g) in a special centrifuge (Medifuge, Silfradent, Italy) to obtain two layers: the lower layer of red blood cells and the upper layer of AFG. The AFG at the top of the tube was collected by means of an injector and transferred to the metal godet. It was held for 15-20 minutes for polymerization. After polymerization occurred, the polymerized AFG in the metal gum was applied to the wound surface in the donor site . No suture or tissue glue was used. Adhesive properties of AFG were utilized.
  Arms: autologous fibrin glue (AFG) group
Biological: i-PRF application on palatinal wound healing — 10 ml venous blood collected from the patient was transferred to the tube without any anticoagulants. Based on G force, collected venous blood were centrifuged at 2300 rpm (about 241 g) in a centrifuge (PC-O2, Process for PRF, Nice, France) for 3 minutes to obtain two layers: The two layers are the lower layer of red blood cells and the upper layer of i-PRF. The i-PRF at the top of the tube was collected with a syringe and transferred to the metal godet. It was held for 20-25 minutes for polymerization. After the polymerization, the polymerized i-PRF was applied to the wound surface in the donor site. No suture or tissue glue was used. Adhesive properties of AFG were utilized.
  Arms: injectable platelet rich fibrin (i-PRF) group
Other: control — no application
  Arms: Control Group

SUMMARY:
Platelet concentrates used in palatal wound healing have been reported to accelerate wound healing and reduce postoperative patient discomfort. The use of elet platelet rich fibrin '(PRF) in the palatal donor site after FGG surgery has been shown to provide significant benefits in terms of wound healing parameters and postoperative comfort. In a study using a platelet rich plasma (PRP) with a different platelet concentration, PRP was found to accelerate wound healing and shorten the healing time. In another study using titanium-prepared platelet rich fibrin (T-PRF) for palatal wound healing, it accelerated the wound healing process and reached the initial level of soft tissue thickness in the donor region at the end of 6 months. In the literature, there are few studies using platelet concentrates in palatal wound healing and only some concentrates (PRP, PRF, T-PRF) are used. The aim of this study is to compare the effects of injectable platelet rich fibrin (i-PRF), which are autologous fibrin glue (AFG) and injectable platelet concentrates, on palatal wound healing. The findings obtained from this study will contribute to the literature in determining the product and method that will provide optimal postoperative patient comfort and wound healing.

DETAILED DESCRIPTION:
Attached gingiva plays an important role in maintaining periodontal health. In the presence of inadequate attached gingiva, periodontal tissue inflammation, root sensitivity, root caries and gingival recessions are caused due to mucogingival stress in the related area and oral hygiene which is not provided adequately. In such cases, inadequate attached gingival width should be increased with mucogingival periodontal plastic surgery.

Free gingival graft (FGG) is accepted as the most commonly used mucogingival procedure in increasing the attached gingival, because of its predictable surgical outcome, simple technique and its application in large areas of operation. In the free gingival graft operation, the recipient bed is prepared in the area with insufficient attached gingiva. Free gingival grafts containing epithelial and connective tissue from the donor area are applied to this recipient bed in appropriate dimensions . Palatal region is the most preferred donor site in terms of anatomical advantage, ideal tissue thickness and wide keratinized band removal. The secondary wound in the donor site after FGG heals in 2-4 weeks and may cause problems that affect patient comfort such as paresthesia, herpetic lesion, mucocele, bleeding and pain in the postoperative period. Different products such as hemostatic agents, low-dose laser treatments, herbal products, ozonated oil, antibacterial / antiseptic agents, bioactive materials and platelet concentrates have been tested to accelerate wound healing and prevent these problems. Studies on the determination of the product and method that provide optimal postoperative patient comfort and wound healing from such products, whose effects on wound healing are known, are ongoing.

Platelet concentrates used in palatal wound healing have been reported to accelerate wound healing and reduce postoperative patient discomfort. The use of elet platelet rich fibrin '(PRF) in the palatal donor site after FGG surgery has been shown to provide significant benefits in terms of wound healing parameters and postoperative comfort. In a study using a platelet rich plasma (PRP) with a different platelet concentration, PRP was found to accelerate wound healing and shorten the healing time. In another study using titanium-prepared platelet rich fibrin (T-PRF) for palatal wound healing, it accelerated the wound healing process and reached the initial level of soft tissue thickness in the donor region at the end of 6 months. In the literature, there are few studies using platelet concentrates in palatal wound healing and only some concentrates (PRP, PRF, T-PRF) are used. The aim of this study is to compare the effects of injectable platelet rich fibrin (i-PRF), which are autologous fibrin glue (AFG) and injectable platelet concentrates, on palatal wound healing. The findings obtained from this study will contribute to the literature in determining the product and method that will provide optimal postoperative patient comfort and wound healing.

In this randomized, controlled clinical study, 36 patients in need of FGG were divided into three groups. AFG (n=12) or i-PRF (n=12) was applied to donor sites and compared to control group (n=12). Wound healing with H2O2 test, VAS, MMS scale and LTH index were evaluated on the 3rd, 7th, 14th day and 1st month. The bleeding status was evaluated on 3rd and 7th days. Palatal tissue thickness was measured at baseline, 1st month and 3rd month.

AFG and i-PRF have positive effects on the healing process by accelerating wound healing and reducing postoperative morbidity.

ELIGIBILITY:
Inclusion Criteria:

* • Patients older than age 18

  * Patients with good oral hygiene
  * Patients who do not use drugs that affect wound healing
  * Patients who are systemically healthy
  * Patients who are non-smokers
  * Patients who do not have coagulation disorder
  * Patients who do not have nausea
  * Patients who are not anti-inflammatory drug allergy sufferers

Exclusion Criteria:

* • Patients who have systematic disorders such as (diabetes, hypertension, radiotherapy, chemotherapy, etc.)

  * Patients who use any medication that may affect wound healing
  * Patients with coagulation disorders
  * Patients who are smokers and alcohol users
  * Patients who are pregnant and breastfeeding
  * Patients with poor oral hygiene
  * Patients who have nausea
  * Patients who are anti-inflammatory drug allergy sufferers
  * Patients who do not attend regular check-ups

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Change of Epithelialization of wound in % at different time points | Epithelialization was evaluated on the 3rd, 7th, 14th day and 1st month.
  Completion of wound epithelialization was evaluated clinically using H2O2 foaming test. After the wound area was dried with gauze, 3% of hydrogen peroxide (H2O2) was applied to the wound with an injector. The result of H2O2 application was evaluated as bubbling within / without palate. The absence of foaming indicates that epithelialization is complete
Change of color, contour and distortion of wound in the total score of scale in numerical at different time points | MMS was evaluated on the 3rd, 7th, 14th day and 1st month.
  The Modified Manchester Scar (MMS) Scale was used to assess the color, contour, and distortion of the wound . The color of the wound was classified as a perfect match (score 0), mild mismatch (score 1), or obvious mismatch (score 2) compared to the neighboring mucosa. The contour of the wound was evaluated as similar (score 0), slightly raised or indented (score 1) and hypertrophic (score 2) when compared to surrounding tissues. Wound distortion was evaluated as no distortion (score 0), mild distortion (score 1) and obvious distortion (score 2) . The sum of the scores in the three categories shows the repair score of the wound, with a total score ranging from 0 to 6, with lower scores indicating better repair.
Change of redness, presence of bleeding, granulation tissue, epithelialization and suppuration in % at different time points | LTH was evaluated on the 3rd, 7th, 14th day and 1st month.
  Wound healing was evaluated using the Landry, Turnbull, Howley (LTH) index, which classifies the healing process according to redness, presence of bleeding, granulation tissue, epithelialization and suppuration. Improvement in this index was scored between 1 (very poor recovery) and 5 (excellent recovery).The sum of the scores shows the repair score of the wound. Evaluation of wound healing process with LTH index was performed on the 3rd, 7th and 14th days and on the 1st and 3rd month controls.

SECONDARY OUTCOMES:
change of Postoperative Pain Evaluation (VAS) in total score of scale in numerical at different time points | VAS was evaluated on the 3rd, 7th, 14th day and 1st month.
  VAS was used for postoperative pain evaluation. On the two ends of a 100 mm line, the definition of 'no pain 'and 'the most severe pain of my life' was written and the patient was asked to mark the appropriate position on this line. The distance from the no pain 'end to the patient's mark was measured in millimeters to determine the patient's pain. Pain assessment was performed on the 3rd, 7th, 14th and 1st month.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA Ö USLU, Asst. Prof., Study Director — Inonu University, Faculty of Dentistry, Department of Periodontics,
Locations (1):
- Inonu University, Faculty of Dentistry, Department of Periodontics,, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No